CLINICAL TRIAL: NCT05610228
Title: Study of the Metabolic Reprogramming of CLL Cells in Ex-vivo Models of the Lymphatic Niche
Brief Title: Study of the Metabolism in the Lymphatic Niche of CLL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Laboimmuno01
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: CLL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA-anticoagulated whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LLC
  Interventions: Other: NO intervention

INTERVENTIONS:
Other: NO intervention — No intervention

SUMMARY:
Chronic lymphoid leukemia (CLL) is the most common adult leukemia that is characterized by a malignant monoclonal accumulation of tumoral and quiescent B cells in the peripheral blood. In advanced stages of the disease (Binet stage C), this population invades the bone marrow (BM) and proliferate into the lymphoid organs that results in widespread adenopathy. Richter's transformation is a most aggressive serious complication of CLL (transformation of the disease into an aggressive lymphoma) detected based on TEP/CT (Positron Emission Tomography/ computerized tomography) that shows highly derived glucose consumption by cancer cells. Clinical data from CLL patients with disease acutisation showed hypermetabolic lymphadenopathy with high standardized uptake value (SUV) whereas there is low grade tracer uptake into BM. We supposed that the tumor microenvironment of the lymphatic niche promotes the proliferation and glycolytic activity of CLL cells which become particularly resistant to treatment. The development of an ex-vivo tumor model that reproduces the microenvironment of the lymph node niche appears essential to identify and validate new therapeutic targets because despite the therapeutic arsenal available some patients still relapse or are refractory to treatment. Our objectives are to i / Characterize this niche of resistance by the development of an ex-vivo tumor model and ii / Evaluate in-vitro the effectiveness of the association of current treatments (RFC, Ibrutinib or Venetoclax) with anti-metabolic therapies (inhibitors of glycolysis) Our lab is developing an ex-vivo models of the lymphatic niche in CLL based on co-cultures of leukemic cells from patients stimulated with CpG ODN and IL2 with primary human lymphatic fibroblasts (HLF) (EC 12PP15). This co-culture has never been described in the literature and allows us to study the lymphatic niche of CLL patients. Lymph node (LN) exploration in CLL requires invasive access and does not bring any additional information in initial diagnosis. Then, we validated our co-culture model using complementary approaches: increased viability, proliferation, and resistance to Ibrutinib, associated with increased production of anti-apoptotic proteins such as MCL1 and BCL2 after 48 hours of co-culture. Secondly, we studied the metabolism in this resistance niche. We find an increased production of lactate and an acute consumption of glucose, associated with a strong metabolic activation detected by SEAHORSE and by the production of glycolysis enzymes such as hexokinase 2. Our study constitutes an original project because it characterized the energy metabolism of the CLL lymphatic niche by developing an original ex-vivo model and enhanced our understanding of the contribution of the specific microenvironment in the dissociation of metabolic activity using SUV max in BM and lymphatic niche. Anti-metabolic therapies are efficient on co-culture CLL cells and could be an alternative for refractory or relapsed patients under current treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom the diagnosis of CLL has been established cytologically and phenotypically (Matutes score)
* Patients over 18 years old
* Patients who have signed the non-objection form
* Untreated patients

Exclusion Criteria:

* Patient with a solid cancer that is progressive or in remission for less than 3 years
* HIV positive patients
* Patients with chronic active hepatitis B or C
* History of allogeneic transplant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLL patient
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Modelisation of a CLL lymphatic niche by creation of an ex-vivo model | 48 months
  Measure of viability and proliferation of CLL cells by annexin PI with multiparameter:
  flow cytometry device, western blot and validation of the model by testing current therapy (Ibrutinib, anti BTK inhibitor)
Study of metabolism in CLL ex-vivo model | 48 months
  Anlayse of metabolism (ECAR and OCR) by seahorse methods , PCR qnd protein Multiparameter analyse
Evaluate in-vitro the effectiveness of the combination of current treatments (RFC, Ibrutinib or Venetoclax) with anti-inflammatory therapies. -metabolic (glycolysis inhibitors) | 48 months
  Viability using multiparameter flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No